CLINICAL TRIAL: NCT06913101
Title: Comparison of Efficacy of Once Weekly Dose of Trelagliptin Versus Once Daily Dose of Vildagliptin on the Levels of HbA1c in Type-2 Diabetes Patients
Brief Title: Comparison of Once-Weekly Trelagliptin vs. Once-Daily Vildagliptin for HbA1c Reduction in Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PNS Hafeez - Naval Hospital (Other Government)
Responsible Party: Principal Investigator, Hamza Ali, Principal Investigator, PNS Hafeez - Naval Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNSHafeez1
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; HbA1c Reduction; Antidiabetic Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Trelagliptin (Experimental): Participants received trelagliptin 100 mg administered orally once weekly before breakfast on the same day of the week.
  Interventions: Drug: Trelagliptin 100 mg
- Group Vildagliptin (Active Comparator): Participants received vildagliptin 50 mg administered orally once daily.
  Interventions: Drug: Vildagliptin 50 mg

INTERVENTIONS:
Drug: Trelagliptin 100 mg — Trelagliptin 100 mg was administered orally once weekly before breakfast on the same day of the week.
  Arms: Group Trelagliptin
Drug: Vildagliptin 50 mg — Vildagliptin 50 mg was administered orally once daily.
  Arms: Group Vildagliptin

SUMMARY:
This randomized controlled trial evaluated the efficacy of once-weekly trelagliptin compared to once-daily vildagliptin in reducing HbA1c levels in patients with type 2 diabetes mellitus (T2DM). A total of 102 participants, aged 30-60 years with HbA1c levels between 7.5% and 9.5%, were enrolled and randomly assigned to either the trelagliptin or vildagliptin group. The primary outcome measured was the percentage of participants achieving an HbA1c level of less than 7% after three months of treatment. Secondary outcomes included the mean reduction in HbA1c levels from baseline. The study aimed to determine whether trelagliptin, with its once-weekly dosing regimen, could improve medication adherence and glycemic control compared to the conventional daily administration of vildagliptin. Data were analyzed using SPSS version 26.0, with independent t-tests and chi-square tests employed for statistical comparisons. Findings from this study contributed to the understanding of the clinical effectiveness of weekly versus daily DPP-4 inhibitors in the management of T2DM.

DETAILED DESCRIPTION:
Before the commencement of the study, ethical approval was obtained from the Institutional Review Board of the hospital. All study procedures adhered strictly to the ethical guidelines of both institutions, ensuring the confidentiality and privacy of all participant data. Potential study participants were provided with detailed information about the study protocols, including the objectives, procedures, potential risks, and benefits of participation. Informed consent was obtained from all participants who met the inclusion criteria and agreed to participate after fully understanding the study details. Participants were diagnosed with type 2 diabetes according to standard diagnostic criteria as per the operational definition. A detailed history was taken to gather basic demographic and clinical data such as age, gender, and comorbidities. Baseline laboratory investigations, including liver function tests (LFTs), renal function tests (RFTs), serum electrolytes, and fundoscopy, were conducted to ensure participants met the selection criteria.

Eligible participants were randomly assigned to one of two treatment groups (Group A or Group B) using a lottery method to ensure equal and unbiased distribution.

Group A received trelagliptin 100 mg once weekly before breakfast on the same day of the week. Group B received vildagliptin 50 mg once daily. Both groups followed the prescribed treatment regimen for a duration of three months. Participants were followed up at three months of treatment. Outcome assessments included monitoring the mean reduction in HbA1c levels and evaluating the efficacy of the treatment, aiming for an HbA1c level of less than 7% after three months of treatment. Data were collected using a data collection proforma.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-60 years.
* Both male and female.
* Diagnosed with type 2 diabetes mellitus.
* HbA1c levels between 7.5% and 9.5% at screening.
* Able to provide informed consent.

Exclusion Criteria:

* Type 1 diabetes mellitus or a history of ketoacidosis.
* Use of insulin or any antidiabetic drugs other than metformin within 3 months prior to the start of the study.
* Significant cardiovascular disease, including recent myocardial infarction (within the last 6 months), unstable angina, or uncontrolled hypertension.
* Chronic kidney disease (stage 3 or worse) or hepatic or pancreatic dysfunction.
* Pregnant or breastfeeding or planning to become pregnant during the study duration.
* Participation in another clinical trial within 30 days prior to enrollment.
* Known hypersensitivity to trelagliptin, vildagliptin, or any components of their formulations.
* Any medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study.
* Participants for whom blood sugar control by insulin preparations is desired (for example, participants with severe ketosis, diabetic coma or precoma, type 1 diabetes mellitus, severe infection, or serious trauma before or after surgery).
* Participants with unstable proliferative diabetic retinopathy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving HbA1c <7% | At 3 months after treatment initiation
  The primary outcome measure was the proportion of participants in each treatment group (trelagliptin vs. vildagliptin) who achieved an HbA1c level of less than 7% after three months of treatment. This outcome assessed the efficacy of once-weekly trelagliptin compared to once-daily vildagliptin in glycemic control among patients with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Mean Reduction in HbA1c Levels | At 3 months after treatment initiation
  The secondary outcome measure was the mean reduction in HbA1c levels from baseline to three months post-treatment in both groups. This outcome evaluated the extent of glycemic improvement achieved with trelagliptin versus vildagliptin.

CONTACTS AND LOCATIONS:
Overall Officials: Hamza Ali, Principal Investigator — PNS Hafeez - Naval Hospital
Locations (1):
- PNS Hafeez - Naval Hospital, Islamabad, Federal Territory, Pakistan

IPD SHARING:
Plan to Share IPD: No